CLINICAL TRIAL: NCT00927485
Title: Use of Curcumin for Treatment of Intestinal Adenomas in Familial Adenomatous Polyposis (FAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marcia R. Cruz-Correa, MD, PhD, Director of Gastrointestinal Oncology, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol A2210108-UPR
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial Adenomatous Polyposis (FAP); Curcumin; Colorectal polyps; Duodenal polyps
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Curcumin; Blood Specimen Collection; Biopsy; Sigmoidoscopy; Gastroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin (Experimental): Curcumin
  Interventions: Drug: Calcumin (Curcumin); Other: Risk Factor Questionnaire; Other: Blood samples; Other: Biopsies (Sigmoidoscopy); Other: Biopsies (Upper endoscopy)
- Placebo (Placebo Comparator): Placebo (sugar pills)
  Interventions: Drug: Calcumin (Curcumin); Other: Risk Factor Questionnaire; Other: Blood samples; Other: Biopsies (Sigmoidoscopy); Other: Biopsies (Upper endoscopy)

INTERVENTIONS:
Drug: Calcumin (Curcumin) — Patients will be randomized to curcumin (3 curcumin pills twice a day for 12 months).
  Other Names: Curcumin
Other: Risk Factor Questionnaire — Questions about current and past lifestyle, health background, and medications. This will take about 20 minutes.
Other: Blood samples — Three tubes of blood at visits 0, 4 and 12 months.
Other: Biopsies (Sigmoidoscopy) — Flexible sigmoidoscopy at baseline and every 4 months for the length of the study (4 months, 8 months, 12 months and 16 months). We will take 2-4 tissue samples of the colon lining by a pinch biopsy.
Other: Biopsies (Upper endoscopy) — Other: Biopsies (Upper endoscopy) Upper endoscopy at baseline and at 12 months. We will take 2-4 tissue samples of the small intestine lining by a pinch biopsy.

SUMMARY:
Familial Adenomatous Polyposis (FAP) is an autosomal dominant disorder characterized by the formation of multiple adenomatous colorectal polyps usually in the teenage years. Virtually, all patients with FAP will develop colorectal cancer on average by the 5th decade of life if prophylactic surgery is not performed. Besides, these individuals must have lifelong cancer surveillance of the remaining colorectum or ileum.

Use of nonsteroidal anti-inflammatory drug (NSAID), such as sulindac, or celecoxib, which selectively inhibits prostaglandin synthesis primarily via the inhibition of cyclogenase-2 (COX-2) have been shown to reduce the incidence and induce regression of adenomas in the rectum of patients with FAP. However, use of NSAIDs and COX-2 inhibitors is associated with significant comorbidity including renal and gastric toxicity and increased risk of vascular events. Therefore, identification of a chemopreventive agent that would have similar efficacy but less toxicity would enhance our ability to treat these patients. Therefore the following specific aim has been proposed:To determine in a randomized, double-blinded, placebo-controlled study the tolerability and efficacy of curcumin to regress intestinal adenomas by measuring duodenal and colorectal/ileal polyp number, and polyp size in patients with FAP.

DETAILED DESCRIPTION:
Patients will be randomized to curcumin (2 curcumin pills twice a day for 12 months) or placebo (2 pills twice a day for 12 months). Besides, blood samples, risk factor questionnaire,and biopsies (upper endoscopy and sigmoidoscopy) will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* 21-85 years with FAP (with an intact colon or who have had surgery)

Exclusion Criteria:

* Mentally incompetent
* Female patients of childbearing age not on effective birth control
* Patients with WBC < 3,500/ml, platelet count < 100,000/ml, BUN > 25mg%, creatinine > 1.5mg%
* Patients unable to stop NSAIDS or aspirin use for the duration of the study
* Malignancy other than nonmelanoma skin cancer
* Active bacterial infection
* Patients with GERD (Gastro esophageal reflux disease)
* Patients with a history of peptic (stomach or duodenal) ulcer disease
* Patients on Warfarin or anti-platelet drugs

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia R. Cruz-Correa, MD. PhD, Principal Investigator — University of Puerto Rico Comprehensive Cancer Center
Locations (1):
- University of Puerto Rico Comprehensive Cancer Center, San Juan, Puerto Rico

REFERENCES:
- [Result] Cruz-Correa M, Hylind LM, Marrero JH, Zahurak ML, Murray-Stewart T, Casero RA Jr, Montgomery EA, Iacobuzio-Donahue C, Brosens LA, Offerhaus GJ, Umar A, Rodriguez LM, Giardiello FM. Efficacy and Safety of Curcumin in Treatment of Intestinal Adenomas in Patients With Familial Adenomatous Polyposis. Gastroenterology. 2018 Sep;155(3):668-673. doi: 10.1053/j.gastro.2018.05.031. Epub 2018 May 23. PMID 29802852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from September 2011 to November 2016 at the Johns Hopkins Hospital and the University of Puerto Rico Medical Sciences Campus. Participants were identified and recruited from the Johns Hopkins Polyposis Registry or from the University of Puerto Rico Familial Colorectal Cancer Registry.
Pre-assignment Details: Absence of effective birth control; pregnancy; WBC < 3500/ml; platelet < 100,000/ml, BUN > 25 mg/dl, Creat > 1.5 mg/dl; malignancy; unwillingness to discontinue NSAIDs; active reflux; hx of peptic ulcer; active bacterial infection; use of warfarin or antiplatelets; allergy to curcumin. 3 month washout period for individuals taking NSAIDs, curcumin, turmeric, aspirin, calcium, vitamin D, green tea or polyphenol E
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 21 | 23
Completed | 15 | 19
Not Completed | 6 | 4
Not completed — Adverse Event | 4 | 2
Not completed — noncompliance, prophylactic surgery, inc | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (1) | 38.7 (1) | 41.6 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Polyps
Description: To determine in a randomized, double-blinded, placebo-controlled study the tolerability and efficacy of curcumin to regress intestinal adenomas by measuring duodenal and colorectal/ileal polyp number in patients with FAP.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: Number of Polyps
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 21 | 23
Number of Polyps | 18.6 [12.1 to 33.1] | 22.6 [9.93 to 27.8]

2. Primary Outcome: Size of Polyps
Description: To determine in a randomized, double-blinded, placebo-controlled study the tolerability and efficacy of curcumin to regress intestinal adenomas by measuring duodenal and colorectal/ileal polyp size in patients with FAP.
Time Frame: 5 years
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 21 | 23
mm | 2.3 [1.8 to 2.8] | 2.1 [1.5 to 2.7]

ADVERSE EVENTS:
Time Frame: Five Years
Arm/Group | Curcumin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 5/21 | 5/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curcumin (N=21) | Placebo (N=23)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No